CLINICAL TRIAL: NCT05198310
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled Study to Assess the Safety, Pharmacokinetics, and Efficacy of KPL-404 in Subjects With Moderate to Severe Active Rheumatoid Arthritis With Inadequate Response or Intolerance to at Least One Biologic Disease-modifying Anti-rheumatic Drug or a Janus Kinase Inhibitor
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Efficacy of KPL-404 in Participants With Rheumatoid Arthritis With Inadequate Response or Intolerance to at Least One Biologic Disease-modifying Anti-rheumatic Drug or a Janus Kinase Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kiniksa Pharmaceuticals International, plc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPL-404-C211; 2022-000169-42 (EudraCT Number)
Record Dates: First submitted 2022-01-03; First posted 2022-01-20 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: inadequate responders; moderate to severe; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 KPL-404 2 mg/kg Every 2 Weeks (q2wk) (Experimental): KPL-404 2 mg/kg subcutaneous (SC) q2wk for 12 weeks
  Interventions: Drug: KPL-404
- Cohort 1 Placebo (Placebo Comparator): Placebo SC q2wk for 12 weeks
  Interventions: Drug: Placebo
- Cohort 2 KPL-404 5 mg/kg q2wk (Experimental): KPL-404 5 mg/kg SC q2wk for 12 weeks
  Interventions: Drug: KPL-404
- Cohort 2 Placebo (Placebo Comparator): Placebo SC q2wk for 12 weeks
  Interventions: Drug: Placebo
- Cohort 3 KPL-404 5 mg/kg qwk (Experimental): KPL-404 5mg/kg SC once weekly (qwk) for 12 weeks
  Interventions: Drug: KPL-404
- Cohort 3 KPL-404 5 mg/kg q2wk (Experimental): KPL-404 5mg/kg SC q2wk with alternating weekly administrations of KPL-404 or placebo SC for 12 weeks
  Interventions: Drug: KPL-404; Drug: Placebo
- Cohort 3 Placebo (Placebo Comparator): Placebo SC qwk for 12 weeks
  Interventions: Drug: Placebo
- Cohort 4 KPL-404 400 mg q4wk (Experimental): KPL-404 SC every 4 weeks (q4wk) for 12 weeks: 600 mg loading dose at baseline followed by 400 mg at Weeks 4 and 8.
  Interventions: Drug: KPL-404
- Cohort 4 Placebo (Placebo Comparator): Placebo SC q4wk for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPL-404 — Humanized monoclonal antibody
  Other Names: abiprubart
  Arms: Cohort 1 KPL-404 2 mg/kg Every 2 Weeks (q2wk); Cohort 2 KPL-404 5 mg/kg q2wk; Cohort 3 KPL-404 5 mg/kg q2wk; Cohort 3 KPL-404 5 mg/kg qwk; Cohort 4 KPL-404 400 mg q4wk
Drug: Placebo — Matching placebo
  Arms: Cohort 1 Placebo; Cohort 2 Placebo; Cohort 3 KPL-404 5 mg/kg q2wk; Cohort 3 Placebo; Cohort 4 Placebo

SUMMARY:
Phase 2 study of the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of KPL-404 in subjects with moderate to severe Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is a 28-week (up to 4-week screening period, 12-week treatment period, and 12-week safety follow-up period), multicenter, randomized, double-blind, placebo-controlled, multiple dose, proof-of-concept study with PK lead-in designed to assess the safety, PK, efficacy and PD of KPL-404 in subjects with moderate to severe, active Rheumatoid Arthritis (RA) who have an inadequate response to or are intolerant to a Janus kinase inhibitor (JAKi) AND/OR at least one biologic disease-modifying anti-rheumatic drug (bDMARD). The objectives of the study are to evaluate safety, efficacy, and PD of KPL-404 compared with placebo across the estimated therapeutic range and to characterize PK across varying dose levels of KPL-404.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 to ≤ 140 kg for all cohorts.
* Diagnosis of RA for ≥ 3 months fulfilling the 2010 American College of Rheumatology (ACR)/European Union League Against Rheumatism (EULAR) classification criteria for RA and that is categorized as ACR RA functional Class 1-3.
* Treated with a biological disease-modifying anti-rheumatic drug (bDMARDs) AND/OR Janus kinase inhibitor (JAKi) therapy for RA for ≥ 3 months and had inadequate response or had to discontinue bDMARD AND/OR JAKi therapy due to intolerance or toxicity, regardless of treatment duration.
* Currently receiving conventional synthetic disease-modifying anti-rheumatic drugs (csDMARD) therapy ≥ 3 months and on a stable dose for ≥ 4 weeks before the first dose of investigational product.

  1. The following csDMARDs are allowed: oral or parenteral methotrexate ([MTX]; 7.5 to 25 mg/week), sulfasalazine (≤ 3000 mg/day), hydroxychloroquine (≤ 400 mg/day), chloroquine (≤ 250 mg/day), and leflunomide (≤ 20 mg/day).
  2. A combination of up to 2 background csDMARDs is allowed, except the combination of MTX and leflunomide.
* Meets all of the following disease activity criteria:

  1. Six or more swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at screening and baseline visits;
  2. Level of high-sensitivity C-reactive protein ≥ 3 mg/L (by central laboratory);
  3. Documented seropositivity for serum Rheumatoid Factor (RF) and/or Anti-citrullinated protein antibody (ACPA) (>ULN) at screening or by prior laboratory evaluation.
* Has completed a locally approved authorized COVID-19 vaccine regimen according to local guidance at least 3 weeks before the first dose of the Investigational Product.
* Must have discontinued all bDMARDs or JAKi prior to the first dose of investigational product. The washout period for bDMARDs or JAKi prior to the first dose of investigational product is specified below. For bDMARDs or JAKi not listed below washout should be at least 5 times the mean elimination half-life of a drug:

  1. ≥ 4 weeks for etanercept;
  2. ≥ 8 weeks for adalimumab, infliximab, certolizumab, golimumab, abatacept, tocilizumab, and sarilumab;
  3. ≥ 1 year for rituximab;
  4. ≥ 2 weeks for JAKi (either investigational or commercially available treatment).
* Voluntarily sign and date an informed consent form approved by independent ethics committee/Institutional Review Board (IRB)

Exclusion Criteria:

* Prior exposure to any other anti-CD40/CD40L agent.
* Inadequate response to 5 or more classes of advanced targeted therapies (bDMARD or tsDMARD; e.g., TNF inhibitors, IL-6 receptor inhibitors, T-cell costimulatory inhibitors, anti-CD-20 antibodies, JAK inhibitors). This does not include prior discontinuation due to drug intolerance.
* Injectable corticosteroids (including intra-articular) or treatment with > 10 mg/day dose oral prednisone or equivalent within 8 weeks prior to randomization.
* History of any arthritis with onset prior to age 16 years or current diagnosis of inflammatory joint disease other than RA (Current diagnosis of secondary Sjogren's syndrome is permitted).
* History of thromboembolic event or a significant risk of future thromboembolic events
* Clinically significant active infection including signs/symptoms suggestive of infection, any significant recurrent or chronic infection, or subjects at a high risk of infection
* History of cancer within the last 5 years from screening, except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured.
* History of any of the following cardiovascular conditions:

  1. Moderate to severe congestive heart failure (New York Heart Association class III or IV);
  2. Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting;
  3. Uncontrolled hypertension as defined by a confirmed systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
* Clinically relevant or significant electrocardiogram (ECG) abnormalities, including ECG with QT interval corrected for heart rate (QTc) > 500 msec.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (19):
  - Carewell Arthritis Center, Apple Valley, California
  - Medvin Clinical Research, Covina, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Medvin Clinical Research, Whittier, California
  - International Medical Research, Daytona Beach, Florida
  - Sweet Hope Research Specialty, Inc., Hialeah, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Millennium Research, Ormond Beach, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Saint Francis Hospital- Memphis, Memphis, Tennessee
  - Arthritis and Rheumatology Research Institute, Allen, Texas
  - Trinity Universal Research Assoc, Carrollton, Texas
  - Arthritis & Osteoporosis Center of Coastal Bend, Corpus Christi, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - DM Clinical Research, Tomball, Texas
  - Rheumatology Clinic of Houston, Tomball, Texas
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Medical center "Artmed" LTD, Plovdiv, Bulgaria
- Czechia (3):
  - Vesalion s.r.o., Ostrava
  - Revmatologicky Utsav, Prague
  - Medical Plus S.R.O., Uherské Hradiště
- Georgia (4):
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - LTD Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
  - JSC Evex Hospitals, Tbilisi
  - LTD Georgian-Dutch Hospital, Tbilisi
- Hungary (6):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Qualiclinic Ltd (Qualiclinic Inc), Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Porcika Klinika, Hódmezővásárhely
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Vita Verum Medical Egeszsegugy, Székesfehérvár
- Poland (5):
  - Centrum Kliniczno-Badawcze, Elblag
  - Silmedic sp. z o.o., Katowice
  - Prywatna Praktyka Lekarska Prof. UM dr hab.med. Pawel Hrycaj, Poznan
  - RCMed Oddzial Sochaczew, Sochaczew
  - Centrum Medyczne Reuma Park, Warsaw
- South Africa (4):
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Jacaranda Hospital, Pretoria, Gauteng
  - Umhlanga Hospital Medical Center, Umhlanga, KwaZulu-Natal
  - Panorama Medical Centre, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1/2 Placebo: Placebo SC q2wk for 12 weeks
  (Per protocol, placebo arms for Cohorts 1 and 2 were combined for analysis.)
- Cohort 3 KPL-404 5 mg/kg Qwk: KPL-404 5 mg/kg SC once weekly (qwk) for 12 weeks
- Cohort 3 KPL-404 5 mg/kg q2wk: KPL-404 5 mg/kg SC q2wk with alternating weekly administrations of KPL-404 or placebo SC for 12 weeks
Period: Overall Study
Arm/Group | Cohort 1 KPL-404 2 mg/kg Every 2 Weeks (q2wk) | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
Started | 6 | 6 | 4 | 27 | 25 | 26 | 31 | 20
Completed | 6 | 5 | 4 | 25 | 25 | 24 | 30 | 17
Not Completed | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 KPL-404 2 mg/kg q2wk: KPL-404 2 mg/kg SC q2wk for 12 weeks
- Cohort 1/2 Placebo: Placebo SC q2wk for 12 weeks
- Cohort 3 KPL-404 5 mg/kg Qwk: KPL-404 5 mg/kg SC qwk for 12 weeks
- Cohort 4 KPL-404 400 mg q4wk: KPL-404 SC q4wk for 12 weeks: 600 mg loading dose at baseline followed by 400 mg at Weeks 4 and 8
- Total: Total of all reporting groups
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo | Total
Number analyzed (Participants) | 6 | 6 | 4 | 27 | 25 | 26 | 31 | 20 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (15.59) | 56.3 (13.29) | 59.8 (13.05) | 58.5 (9.68) | 60.0 (10.10) | 57.6 (9.90) | 58.8 (9.45) | 58.3 (11.81) | 58.5 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 22 | 20 | 24 | 25 | 15 | 120
  Male | 1 | 1 | 0 | 5 | 5 | 2 | 6 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 2 | 2 | 3 | 6 | 5 | 1 | 24
  Not Hispanic or Latino | 5 | 2 | 2 | 25 | 22 | 20 | 26 | 19 | 121
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2 | 2 | 3 | 1 | 10
  White | 5 | 6 | 4 | 25 | 23 | 24 | 26 | 17 | 130
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE): any untoward medical occurrence, which does not necessarily have a causal relationship with this treatment. Serious AE (SAE): AE that: results in death; is immediately life-threatening; requires in-patient hospitalization/prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital abnormality/birth defect; is an important medical event. TEAEs: AEs not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug during treatment period. AE severity: mild (Grade [Gr] 1); moderate (Gr 2); severe (Gr 3); potentially life threatening (Gr 4); death (Gr 5). AEs of special interest: thrombosis, serious infection, serious and non-serious bacterial infections, eye disorders, and anaphylaxis/hypersensitivity reactions.
Time Frame: From first dose of study drug to 24 weeks
Population: Safety Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 KPL-404 2 mg/kg q2wk: KPL-404 2 mg/kg SC every 2 q2wk for 12 weeks
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo
Number analyzed (Participants) | 6 | 6 | 4
Participants
  TEAEs | 2 | 2 | 3
  Drug-related TEAEs | 1 | 1 | 1
  TEAEs by maximum severity | 2 | 2 | 3
  Maximum Severity = Mild | 1 | 1 | 1
  Maximum Severity = Moderate | 1 | 1 | 2
  Maximum Severity = Severe | 0 | 0 | 0
  Maximum Severity = Potentially life threatening | 0 | 0 | 0
  Maximum Severity = Fatal | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0
  Drug-related SAEs | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0
  TEAEs leading to dose interruption | 1 | 1 | 0
  TEAEs leading to treatment discontinuation | 0 | 0 | 0
  TEAEs of special interest | 0 | 0 | 0
  Injection site reactions | 0 | 1 | 0

2. Primary Outcome: Cohorts 1 and 2: Maximum Serum Concentration (Cmax)
Time Frame: Days 1 (Dose 1) and 57 (Dose 4)
Population: Participants treated with KPL-404, with an evaluable PK sample at given time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk
Number analyzed (Participants) | 5 | 6
µg/mL
  Day 1 | 7.57 (7.52) | 28.0 (13.5)
  Day 57: number analyzed (Participants) | 3 | 6
  Day 57 | 17.8 (13.9) | 68.3 (25.1)

3. Primary Outcome: Cohorts 1 and 2: Area Under the Serum Concentration-time Curve From Time of Administration to the End of the Dosing Interval, (AUCtau)
Time Frame: Days 1 (Dose 1) and 57 (Dose 4)
Population: Participants treated with KPL-404, with an evaluable PK sample at given time point.
Measure: Mean (Standard Deviation); unit: µg·day/mL
Groups:
- Cohort 1 KPL-404: KPL-404 2 mg/kg SC q2wk for 12 weeks
- Cohort 2 KPL-404: KPL-404 5 mg/kg SC q2wk for 12 weeks
Arm/Group | Cohort 1 KPL-404 | Cohort 2 KPL-404
Number analyzed (Participants) | 5 | 6
µg·day/mL
  Day 1 | 59.0 (51.1) | 303 (148)
  Day 57: number analyzed (Participants) | 3 | 6
  Day 57 | 162 (114) | 810 (290)

4. Primary Outcome: Cohort 3 and 4: Change From Baseline in Disease Activity Score of 28 Joints Using C-reactive Protein (DAS28-CRP) at Week 12
Description: DAS28 is a measure based on assessment of 28 joints for tenderness and swelling (tender and swollen joint counts). DAS28-CRP is derived using differential weighting given to 4 components: tender joint count (range: 0-28), swollen joint count (range: 0-28), patient global assessment (recorded on a visual analog scale [VAS] scale of 0-100 mm), and CRP (milligram per liter). DAS28-CRP score ranges from 0 to 9.4. The lower the DAS28-CRP score is, the better the participant has response (remission = score < 2.6, low disease activity = score < 3.2). A negative value in change from BL indicates an improvement.
Time Frame: Baseline, Week 12
Population: Modified Intent-to-Treat (mITT) population: All randomized participants who received at least one dose of study drug and who had at least one post-baseline assessment for the primary efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
Number analyzed (Participants) | 27 | 25 | 26 | 31 | 20
score on a scale | -2.17 (0.216) | -1.96 (0.220) | -1.61 (0.218) | -1.87 (0.331) | -1.30 (0.338)
Statistical Analysis 1: Comparison: Cohort 3 KPL-404 5 mg/kg Qwk vs Cohort 3 Placebo; Test type: Superiority; p = 0.0470, ANCOVA — Analyzed using ANCOVA model with baseline value and stratification factor (≤1 vs. ≥2 classes of advanced targeted therapies) as covariates; LS Mean Difference = -0.57, 95% CI 2-sided [-1.13 to -0.01], Standard Error of Mean 0.281
Statistical Analysis 2: Comparison: Cohort 3 KPL-404 5 mg/kg q2wk vs Cohort 3 Placebo; Test type: Superiority; p = 0.2124, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.36, 95% CI 2-sided [-0.92 to 0.21], Standard Error of Mean 0.282
Statistical Analysis 3: Comparison: Cohort 4 KPL-404 400 mg q4wk vs Cohort 4 Placebo; Test type: Superiority; p = 0.1091, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.58, 95% CI 2-sided [-1.28 to 0.13], Standard Error of Mean 0.352

5. Secondary Outcome: Cohorts 1 and 2: Change From Baseline in DAS28-CRP at Week 12
Description: as for outcome 4
Time Frame: Baseline, Week 12
Population: mITT Population: All randomized participants who received at least one dose of study drug and who had at least one post-baseline assessment for the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo
Number analyzed (Participants) | 6 | 6 | 4
score on a scale | -3.16 (1.130) | -3.44 (1.450) | -1.09 (1.373)
Statistical Analysis 1: Comparison: Cohort 1 KPL-404 2 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 0.0312, t-test
Statistical Analysis 2: Comparison: Cohort 2 KPL-404 5 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 0.0338, t-test

6. Secondary Outcome: Cohorts 3 and 4: Number of Participants With TEAEs
Description: as for outcome 1
Time Frame: From first dose of study drug to 24 weeks
Population: Safety Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
Number analyzed (Participants) | 27 | 25 | 26 | 31 | 20
Participants
  TEAEs | 12 | 6 | 8 | 9 | 8
  Drug-related TEAEs | 2 | 2 | 2 | 3 | 1
  TEAEs by maximum severity | 12 | 6 | 8 | 9 | 8
  Maximum Severity = Mild | 8 | 3 | 4 | 4 | 5
  Maximum Severity = Moderate | 4 | 3 | 4 | 5 | 3
  Maximum Severity = Severe | 0 | 0 | 0 | 0 | 0
  Maximum Severity = Potentially life threatening | 0 | 0 | 0 | 0 | 0
  Maximum Severity = Fatal | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 1 | 0 | 0 | 0 | 0
  Drug-related SAEs | 0 | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0
  TEAEs leading to dose interruption | 1 | 0 | 1 | 0 | 0
  TEAEs leading to treatment discontinuation | 0 | 0 | 0 | 1 | 1
  TEAEs of special interest | 1 | 1 | 0 | 1 | 2
  Injection site reactions | 1 | 1 | 0 | 2 | 0

7. Secondary Outcome: Cohort 3 and 4: Cmax
Time Frame: Days 1 (Dose 1) and 57 (Dose 4 or 8)
Population: Participants treated with KPL-404, with an evaluable PK sample at given time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Cohort 3 KPL-404 5 mg/kg Qwk: KPL-404 5mg/kg SC qwk for 12 weeks
Arm/Group | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 4 KPL-404 400 mg q4wk
Number analyzed (Participants) | 27 | 25 | 30
µg/mL
  Day 1 | 27.1 (11.0) | 29.4 (10.3) | 48.5 (18.2)
  Day 57: number analyzed (Participants) | 22 | 25 | 27
  Day 57 | 145 (41.0) | 70.9 (21.5) | 45.6 (21.4)

8. Secondary Outcome: Cohort 3 and 4: AUCtau
Time Frame: Days 1 (Dose 1) and 57 (Dose 4 or 8)
Population: Participants treated with KPL-404, with an evaluable PK sample at given time point.
Measure: Mean (Standard Deviation); unit: µg·day/mL
Arm/Group | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 4 KPL-404 400 mg q4wk
Number analyzed (Participants) | 27 | 25 | 30
µg·day/mL
  Day 1 | 139 (63.4) | 310 (105) | 873 (363)
  Day 57: number analyzed (Participants) | 22 | 25 | 27
  Day 57 | 975 (291) | 849 (267) | 843 (466)

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: An ACR20 response is defined as at least a 20% improvement in both tender joint count (TJC) and swollen joint count (SJC), and at least a 20% improvement in three of the following five criteria: patient global assessment (PGA), physician global assessment (PhGA), functional ability measure [Health Assessment Questionnaire (HAQ)], patient's assessment of pain (visual analog scale; VAS) and C-reactive protein (CRP).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 6 | 4 | 27 | 25 | 26 | 31 | 20
percentage of participants | 100 | 83.3 | 25.0 | 74.1 | 60.0 | 50.0 | 80.6 | 40.0
Statistical Analysis 1: Comparison: Cohort 1 KPL-404 2 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 0.0333, Fisher exact test
Statistical Analysis 2: Comparison: Cohort 2 KPL-404 5 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 0.1905, Fisher exact test
Statistical Analysis 3: Comparison: Cohort 3 KPL-404 5 mg/kg Qwk vs Cohort 3 Placebo; Test type: Superiority; p = 0.0716, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.95, 95% CI 2-sided [0.90 to 9.65]
Statistical Analysis 4: Comparison: Cohort 3 KPL-404 5 mg/kg q2wk vs Cohort 3 Placebo; Test type: Superiority; p = 0.4710, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.50 to 4.67]
Statistical Analysis 5: Comparison: Cohort 4 KPL-404 400 mg q4wk vs Cohort 4 Placebo; Test type: Superiority; p = 0.0057, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.09, 95% CI 2-sided [1.62 to 22.88]

10. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Week 12
Description: An ACR50 response is defined as at least a 50% improvement in both tender joint count (TJC) and swollen joint count (SJC), and at least a 50% improvement in three of the following five criteria: patient global assessment (PGA), physician global assessment (PhGA), functional ability measure [Health Assessment Questionnaire (HAQ)], patient's assessment of pain (visual analog scale; VAS) and C-reactive protein (CRP).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 6 | 4 | 27 | 25 | 26 | 31 | 20
percentage of participants | 66.7 | 16.7 | 0 | 33.3 | 36.0 | 23.1 | 32.3 | 30.0
Statistical Analysis 1: Comparison: Cohort 1 KPL-404 2 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 0.0762, Fisher exact test
Statistical Analysis 2: Comparison: Cohort 2 KPL-404 5 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 1.000, Fisher exact test
Statistical Analysis 3: Comparison: Cohort 3 KPL-404 5 mg/kg Qwk vs Cohort 3 Placebo; Test type: Superiority; p = 0.4172, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.49 to 5.62]
Statistical Analysis 4: Comparison: Cohort 3 KPL-404 5 mg/kg q2wk vs Cohort 3 Placebo; Test type: Superiority; p = 0.3144, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.55 to 6.45]
Statistical Analysis 5: Comparison: Cohort 4 KPL-404 400 mg q4wk vs Cohort 4 Placebo; Test type: Superiority; p = 0.9560, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.28 to 3.39]

11. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 12
Description: An ACR70 response is defined as at least a 70% improvement in both tender joint count (TJC) and swollen joint count (SJC), and at least a 70% improvement in three of the following five criteria: patient global assessment (PGA), physician global assessment (PhGA), functional ability measure [Health Assessment Questionnaire (HAQ)], patient's assessment of pain (visual analog scale; VAS) and C-reactive protein (CRP).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
Number analyzed (Participants) | 6 | 6 | 4 | 27 | 25 | 26 | 31 | 20
percentage of participants | 33.3 | 16.7 | 0 | 7.4 | 20.0 | 3.8 | 9.7 | 25.0
Statistical Analysis 1: Comparison: Cohort 1 KPL-404 2 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 0.4667, Fisher exact test
Statistical Analysis 2: Comparison: Cohort 2 KPL-404 5 mg/kg q2wk vs Cohort 1/2 Placebo; Test type: Superiority; p = 1.0000, Fisher exact test
Statistical Analysis 3: Comparison: Cohort 3 KPL-404 5 mg/kg Qwk vs Cohort 3 Placebo; Test type: Superiority; p = 0.5789, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.17 to 22.30]
Statistical Analysis 4: Comparison: Cohort 3 KPL-404 5 mg/kg q2wk vs Cohort 3 Placebo; Test type: Superiority; p = 0.0799, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.12, 95% CI 2-sided [0.62 to 60.10]
Statistical Analysis 5: Comparison: Cohort 4 KPL-404 400 mg q4wk vs Cohort 4 Placebo; Test type: Superiority; p = 0.1034, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.06 to 1.35]

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | Cohort 1 KPL-404 2 mg/kg q2wk | Cohort 2 KPL-404 5 mg/kg q2wk | Cohort 1/2 Placebo | Cohort 3 KPL-404 5 mg/kg Qwk | Cohort 3 KPL-404 5 mg/kg q2wk | Cohort 3 Placebo | Cohort 4 KPL-404 400 mg q4wk | Cohort 4 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/27 | 0/25 | 0/26 | 0/31 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 1/27 | 0/25 | 1/26 | 0/31 | 0/20
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 3/4 | 10/27 | 8/25 | 8/26 | 10/31 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 KPL-404 2 mg/kg q2wk (N=6) | Cohort 2 KPL-404 5 mg/kg q2wk (N=6) | Cohort 1/2 Placebo (N=4) | Cohort 3 KPL-404 5 mg/kg Qwk (N=27) | Cohort 3 KPL-404 5 mg/kg q2wk (N=25) | Cohort 3 Placebo (N=26) | Cohort 4 KPL-404 400 mg q4wk (N=31) | Cohort 4 Placebo (N=20)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 KPL-404 2 mg/kg q2wk (N=6) | Cohort 2 KPL-404 5 mg/kg q2wk (N=6) | Cohort 1/2 Placebo (N=4) | Cohort 3 KPL-404 5 mg/kg Qwk (N=27) | Cohort 3 KPL-404 5 mg/kg q2wk (N=25) | Cohort 3 Placebo (N=26) | Cohort 4 KPL-404 400 mg q4wk (N=31) | Cohort 4 Placebo (N=20)
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 2 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publish before a first multi-center publication by Sponsor. Before submission, Sponsor has 60 days to review any manuscript and 30 days to review any poster, abstract or any other materials. If Sponsor requests in writing, Investigator shall withhold disclosure for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT05198310/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT05198310/SAP_001.pdf